CLINICAL TRIAL: NCT03554681
Title: Prospective Validation of Prediction Algorithms for Preeclampsia in the First-trimester of Pregnancy
Brief Title: Prediction of Preeclampsia (PE) at 11-13 Week
Status: Completed | Type: Observational
Sponsor: Chiu Yee Liona Poon (Other)
Responsible Party: Sponsor-Investigator, Chiu Yee Liona Poon, Associate Professor (Clinical), Chinese University of Hong Kong
Organization: Chinese University of Hong Kong (Other)
Other Study IDs: 2016.152
Record Dates: First submitted 2018-05-09; First posted 2018-06-13 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Pre-Eclampsia
Keywords: Bayes Model
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — An additional blood 5ml sample, if agreed to by the study participant, for recovery of plasma for future research will be taken and archived at -80℃.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an international multicentre prospective cohort study to validate the Bayes theorem based algorithms for the screening of pre-eclampsia (PE) in the first-trimester of pregnancy.

DETAILED DESCRIPTION:
The investigators have previously constructed Bayes model in the first-trimester which combines maternal characteristics and medical history (Mat-CH) together with mean arterial pressure (MAP), uterine artery pulsatility index (PI), and serum placental growth factor (PlGF) with a plan to assess the predictive performance.

The reference standards will be PE defined according to the International Society for the Study of Hypertension in Pregnancy and the American College of Obstetricians and Gynecologists. The systolic blood pressure should be >140 mm Hg and/or the diastolic blood pressure should be >90 mmHg on at least two occasions four hours apart developing after 20 weeks' gestation in previously normotensive women and there should be proteinuria (>300 mg in 24 hours or two readings of at >2+ on dipstick analysis of midstream or catheter urine specimens if no 24-hour collection is available). In the absence of proteinuria, new onset of any of the following systemic findings: a) thrombocytopaenia (platelet counts <100,000 µL); b) renal insufficiency (creatinine >1.1 mg/dL or 2-fold increase in creatinine in the absence of underlying renal disease); c) abnormal liver function (ie, hepatic transaminase levels twice normal); d) pulmonary oedema; or e) cerebral or visual symptoms. Preterm-PE is PE that requires delivery before 37 weeks' gestation. If a participant fulfills the criteria for PE by one definition and not the other she will be considered to have developed PE.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Singleton pregnancy
* Live fetus
* Provide Informed and written consent in the official language of the country

Exclusion Criteria:

* Unable to provide written Informed consent learning difficulties or serious mental illness or an inability to understand spoken and written the official language of the country.
* Multiple Pregnancy
* Non-viable fetus (missed spontaneous abortion or stillbirth)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible women attending for their hospital visit at 11-13 weeks will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 10935 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
The false positive and true positive frequencies for screening for PE using the Bayes theorem based methods | At delivery

SECONDARY OUTCOMES:
The false positive and true positive frequencies for screening of delivery of all-Small for Gestational Age (SGA) neonates and preterm-SGA neonates (delivery before 37 weeks), with or without PE | At delivery

CONTACTS AND LOCATIONS:
Overall Officials: Liona CY Poon, Principal Investigator — Chinese University of Hong Kong
Locations (14):
- China (2):
  - First Affiliated Hospital of Kunming Medical University, Kunming
  - Nanjing Drum Tower Hospital, Nanjing
- Hong Kong (2):
  - Kwong Wah Hospital, Hong Kong
  - Prince of Wales Hospital, Hong Kong
- Mediscan Chennai, Chennai, Tamil Nadu, India
- Japan (4):
  - Toyama University Hospital, Toyama, Toyama
  - Clinical Research Institute of Fetal Medicine PMC, Osaka
  - Affiliated hospitals within The Japan Society for the Study of Hypertension in Pregnancy (JSSHP), Tokyo
  - Showa University Hospital, Tokyo
- Singapore (2):
  - KK Women's and Children's Hospital, Singapore
  - National University Hospital, Singapore
- Taipei Chang Gung Memorial Hospital, Taipei, Taiwan
- Thailand (2):
  - Chulalongkorn University Bangkok, Bangkok
  - Siriraj Hospital, Bangkok

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] National Collaborating Centre for Women's and Children's Health (UK). Hypertension in Pregnancy: The Management of Hypertensive Disorders During Pregnancy. London: RCOG Press; 2010 Aug. Available from http://www.ncbi.nlm.nih.gov/books/NBK62652/ PMID 22220321
- [Background] Askie LM, Duley L, Henderson-Smart DJ, Stewart LA; PARIS Collaborative Group. Antiplatelet agents for prevention of pre-eclampsia: a meta-analysis of individual patient data. Lancet. 2007 May 26;369(9575):1791-1798. doi: 10.1016/S0140-6736(07)60712-0. PMID 17512048
- [Background] Bujold E, Roberge S, Lacasse Y, Bureau M, Audibert F, Marcoux S, Forest JC, Giguere Y. Prevention of preeclampsia and intrauterine growth restriction with aspirin started in early pregnancy: a meta-analysis. Obstet Gynecol. 2010 Aug;116(2 Pt 1):402-414. doi: 10.1097/AOG.0b013e3181e9322a. PMID 20664402
- [Background] Roberge S, Villa P, Nicolaides K, Giguere Y, Vainio M, Bakthi A, Ebrashy A, Bujold E. Early administration of low-dose aspirin for the prevention of preterm and term preeclampsia: a systematic review and meta-analysis. Fetal Diagn Ther. 2012;31(3):141-6. doi: 10.1159/000336662. Epub 2012 Mar 21. PMID 22441437
- [Background] Roberge S, Giguere Y, Villa P, Nicolaides K, Vainio M, Forest JC, von Dadelszen P, Vaiman D, Tapp S, Bujold E. Early administration of low-dose aspirin for the prevention of severe and mild preeclampsia: a systematic review and meta-analysis. Am J Perinatol. 2012 Aug;29(7):551-6. doi: 10.1055/s-0032-1310527. Epub 2012 Apr 11. PMID 22495898
- [Background] Wright D, Syngelaki A, Akolekar R, Poon LC, Nicolaides KH. Competing risks model in screening for preeclampsia by maternal characteristics and medical history. Am J Obstet Gynecol. 2015 Jul;213(1):62.e1-62.e10. doi: 10.1016/j.ajog.2015.02.018. Epub 2015 Feb 25. PMID 25724400
- [Background] O'Gorman N, Wright D, Syngelaki A, Akolekar R, Wright A, Poon LC, Nicolaides KH. Competing risks model in screening for preeclampsia by maternal factors and biomarkers at 11-13 weeks gestation. Am J Obstet Gynecol. 2016 Jan;214(1):103.e1-103.e12. doi: 10.1016/j.ajog.2015.08.034. Epub 2015 Aug 19. PMID 26297382
- [Background] Gallo DM, Wright D, Casanova C, Campanero M, Nicolaides KH. Competing risks model in screening for preeclampsia by maternal factors and biomarkers at 19-24 weeks' gestation. Am J Obstet Gynecol. 2016 May;214(5):619.e1-619.e17. doi: 10.1016/j.ajog.2015.11.016. Epub 2015 Nov 25. PMID 26627730
- [Background] Tsiakkas A, Saiid Y, Wright A, Wright D, Nicolaides KH. Competing risks model in screening for preeclampsia by maternal factors and biomarkers at 30-34 weeks' gestation. Am J Obstet Gynecol. 2016 Jul;215(1):87.e1-87.e17. doi: 10.1016/j.ajog.2016.02.016. Epub 2016 Feb 12. PMID 26875953
- [Background] Andrietti S, Silva M, Wright A, Wright D, Nicolaides KH. Competing-risks model in screening for pre-eclampsia by maternal factors and biomarkers at 35-37 weeks' gestation. Ultrasound Obstet Gynecol. 2016 Jul;48(1):72-9. doi: 10.1002/uog.15812. Epub 2016 May 30. PMID 26566592
- [Background] Brown MA, Lindheimer MD, de Swiet M, Van Assche A, Moutquin JM. The classification and diagnosis of the hypertensive disorders of pregnancy: statement from the International Society for the Study of Hypertension in Pregnancy (ISSHP). Hypertens Pregnancy. 2001;20(1):IX-XIV. doi: 10.1081/PRG-100104165. No abstract available. PMID 12044323
- [Background] Hypertension in pregnancy. Report of the American College of Obstetricians and Gynecologists' Task Force on Hypertension in Pregnancy. Obstet Gynecol. 2013 Nov;122(5):1122-1131. doi: 10.1097/01.AOG.0000437382.03963.88. No abstract available. PMID 24150027
- [Background] Snijders RJ, Nicolaides KH. Fetal biometry at 14-40 weeks' gestation. Ultrasound Obstet Gynecol. 1994 Jan 1;4(1):34-48. doi: 10.1046/j.1469-0705.1994.04010034.x. PMID 12797224
- [Background] Acharya G, Wilsgaard T, Berntsen GK, Maltau JM, Kiserud T. Reference ranges for serial measurements of umbilical artery Doppler indices in the second half of pregnancy. Am J Obstet Gynecol. 2005 Mar;192(3):937-44. doi: 10.1016/j.ajog.2004.09.019. PMID 15746695
- [Background] Vyas S, Campbell S, Bower S, Nicolaides KH. Maternal abdominal pressure alters fetal cerebral blood flow. Br J Obstet Gynaecol. 1990 Aug;97(8):740-2. doi: 10.1111/j.1471-0528.1990.tb16250.x. No abstract available. PMID 2205291